CLINICAL TRIAL: NCT01986894
Title: A Phase 1, Double-blind, Four Period Crossover Study to Investigate the Effects of Pomalidomide (CC 4047) on the QT Interval in Healthy Male Subjects
Brief Title: A Phase 1 QT Study in Healthy Male Subjects
Acronym: QT/QTc
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CC-4047-CP-010
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Clinical Pharmacology, Healthy Volunteer Study
Keywords: TQT; Pharmacokinetic; Healthy
MeSH Terms: interventions — pomalidomide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (placebo) (Placebo Comparator): Five placebo capsules matching the appearance of the 4 mg pomalidomide capsule will be administered orally on the morning of Day 1
  Interventions: Drug: Placebo
- Treatment 2 (4 mg pomalidomide) (Experimental): Five capsules (one 4 mg pomalidomide capsule and four placebo capsules matching the appearance of the 4 mg pomalidomide capsule) will be administered orally on the morning of Day 1
  Interventions: Drug: Pomalidomide
- Treatment 3 (20 mg pomalidomide) (Experimental): Five 4 mg pomalidomide capsules will be administered orally on the morning of Day 1
  Interventions: Drug: Pomalidomide
- Treatment 4 (moxifloxacin) (Active Comparator): One 400 mg moxifloxacin tablet (AVELOX®, moxifloxacin hydrochloride, Bayer Pharmaceuticals Corporation) will be administered orally on the morning of Day 1
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Placebo — Single oral dose of Placebo
  Arms: Treatment 1 (placebo)
Drug: Pomalidomide — Single oral dose of 4 mg pomalidomide
  Other Names: POMALYST®
  Arms: Treatment 2 (4 mg pomalidomide)
Drug: Pomalidomide — Single oral dose of 20 mg pomalidomide
  Other Names: POMALYST®
  Arms: Treatment 3 (20 mg pomalidomide)
Drug: Moxifloxacin — Single oral dose of 400 mg moxifloxacin tablet
  Other Names: AVELOX®
  Arms: Treatment 4 (moxifloxacin)

SUMMARY:
This is a single-center, randomized, double-blind crossover study with four treatments, four periods and four sequences to investigate the effects of orally administered pomalidomide on QT interval. The study will be conducted in healthy male subjects. Pomalidomide (clinically indicated dose for multiple myeloma [MM] as per the United States Package Insert [USPI] of 4 mg and supratherapeutic dose of 20 mg) and placebo treatments will be double-blinded. Moxifloxacin (positive control) will be administered in an open-label fashion to determine the sensitivity of the assay. The core electrocardiogram (ECG) laboratory and ECG readers will be blinded to all study treatments and sequences.

DETAILED DESCRIPTION:
A total of 72 male subjects will be randomized and enrolled, with 18 subjects assigned to each treatment sequence. For each treatment sequence, each subject will participate in a screening phase, four baseline phases, four treatment periods and a follow up visit. Within 28 days prior to Period 1 dosing, subjects will sign an informed consent document (ICD) and undergo screening procedures to confirm eligibility. Qualifying subjects will return to the clinical site on Day -2 of Period 1 to begin baseline assessments, and will be domiciled at the clinical site from Day -2 to Day 2 of Period 1. For all remaining study periods, subjects will return to the clinical site on Day -1 to begin baseline assessments, and will be domiciled at the clinical site from Day -1 to Day 2. Subjects will be assigned randomly to one of four treatment sequences and will receive a single dose of the assigned treatment on Day 1 of each study period. There will be a minimum of 7 days and no more than 14 days between each dose.

Subjects will begin an overnight fast of at least 8 hours prior to the start of continuous Holter monitoring on Day 1 (and Day 1 in Period 1). On the morning of Day 1 (and Day -1 in Period 1), continuous Holter monitoring for approximately 24 hours will be performed. Triplicate ECGs will be extracted for analysis at specific predose and postdose timepoints (or equivalent times on Day -1 of Period 1). Blood samples will be collected at pre specified timepoints for pharmacokinetic (PK) and clinical laboratory assessments. Safety will be monitored throughout the study.

During each study period, subjects will be discharged from the clinical site on Day 2 upon satisfactory safety review and completion of the required study procedures. A safety follow up will be conducted by telephone 5 to 7 days following discharge in Period 4. In the event that a subject discontinues from the study, an early termination visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must understand and voluntarily sign a written informed consent (ICD) prior to any study related procedures being performed.

  2. Must be able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules 3. Healthy male of any race between 18 to 50 years of age (inclusive) at the time of signing the ICD, and in good health as determined by a physical exam (P)E.

  4. Must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential (FCBP) while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.
* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Period abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception.

  5. Must have a body-mass index (BMI) between 18 and 30 kg/m2 (inclusive). 6. Clinical laboratory tests must be within normal limits or acceptable to the Investigator.

  7. Subject must be afebrile, with supine systolic blood pressure (BP): 90 to 140 mmHg, supine diastolic BP: 60 to 90 mmHg, and pulse rate (PR): 40 to 110 bpm.

At screening: After the supine measurements, when BP and pulse rate are measured again after 5 minutes of standing, there shall be no more than a 20 mmHg drop in systolic BP or no more than a 10 mmHg drop in diastolic BP and/or no more than a 20 bpm increase in pulse rate associated with clinical manifestation of postural hypotension.

8. Must have a normal or clinically acceptable 12-lead electrocardiogram (ECG) at screening; must have a QTcF value ≤ 430 msec.

9. Must agree to refrain from donating sperm or semen while participating in this study and for at least 28 days following the last dose of study drug.

10. Must agree to refrain from donating blood or plasma (other than for this study) while participating in this study and for at least 28 days following the last dose of study drug.

Exclusion Criteria:

* 1. History of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular (including hypertension, atherosclerosis, heart failure, supraventricular or ventricular arrhythmias and stroke [Cerebral Vascular Accident (CVA)] or transient ischemic attack [TIA]), psychological, pulmonary (including asthma and chronic obstructive pulmonary disease [COPD], treated or not treated), metabolic, endocrine, hematological, allergic disease, drug allergies, known hypersensitivity to a member of the class of IMiDs®, known hypersensitivity to moxifloxacin or other major disorders.

  2. Any condition which places the subject at unacceptable risk if he was to participate in the study, or confounds the ability to interpret data from the study.

  3. Have a first degree relative (parent, sibling, child) with Long QT Syndrome. 4. A hemoglobin level of less than 12.0 g/dL. 5. Abnormal Electrocardiogram (ECG) findings as follows:
  * Heart rate < 40 or > 110 bpm, after resting in the supine position for 5 minutes;
  * Pulse rate (PR) interval > 220 msec;
  * QRS interval > 120 including any degree of bundle branch block;
  * QTcF < 300 or > 430 msec;
  * Evidence of pre-excitation (e.g., Wolfe-Parkinson-White syndrome);
  * Cardiac pacemaker;
  * Atrial fibrillation / flutter. 6. QRS and/or T wave that the Investigator judges to be unfavorable for consistently accurate QT measurements (e.g., indistinct QRS onset, low amplitude T wave, inverted or terminally inverted T wave, merged T/U waves, indistinct T wave offset, or prominent U wave that affects QT measurement).

    7. Neuromuscular artifact that cannot readily be eliminated. 8. Subjects with hypokalemia and/or hypomagnesemia condition. 9. Used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of the first dose administration, unless sponsor agreement is obtained.

    10. Used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration, unless sponsor agreement is obtained.

    11. Has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), e.g., bariatric procedure. Appendectomy and cholecystectomy are acceptable.

    12. Donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.

    13. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or positive drug test reflecting consumption of illicit drugs.

    14. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before dosing, or positive alcohol screen.

    15. Known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HbsAg) or hepatitis C virus antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

    16. Exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).

    17. Cotinine level at screening or on Day 2 of Period 1 indicates subject is a moderate or heavy smoker.

    18. History of autonomic dysfunction (e.g., history of fainting or orthostatic hypotension).

    19. Subjects who are part of the clinical staff personnel or family members of the clinical site staff.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
Time matched, baseline corrected change from placebo of QTcF | From before dosing until 23 hours after dosing
  To evaluate the effect of pomalidomide on the time matched changes from placebo in the baseline adjusted QT interval of the electrocardiogram (ECG) using the Fridericia correction method (QTcF)
Categorical analyses on ECG intervals and changes in ECG morphology | From before dosing until 23 hours after dosing

SECONDARY OUTCOMES:
Time matched, baseline corrected changes from placebo of other ECG intervals (RR, PR, QRS) and categorical analyses on ECG intervals and changes in ECG morphology | From before dosing until 23 hours after dosing
  To evaluate the change from placebo in selected ECG parameters (heart rate, PR interval, QRS interval, uncorrected QT interval and morphological patterns) following pomalidomide treatment
Safety | 2 months (from screening visit until end of study
  To assess the safety and tolerability of single oral doses of pomalidomide
Pharmacokinetics - Cmax | From before dosing until 32 hours after dosing
  Maximum observed plasma concentration
Pharmacokinetics - Tmax | From before dosing until 32 hours after dosing
  Time to Cmax
Pharmacokinetics - AUCinf | From before dosing until 32 hours after dosing
  Area under the plasma concentration time curve from time zero extrapolated to infinity
Pharmacokinetics - AUCt | From before dosing until 32 hours after dosing
  Area under the plasma concentration time curve from time zero to the last quantifiable concentration
Pharmacokinetics - t1/2 | From before dosing until 32 hours after dosing
  Terminal phase elimination half-life
Pharmacokinetics - CL/F | From before dosing until 32 hours after dosing
  Apparent total plasma clearance when dosed orally
Pharmacokinetics - Vz/F | From before dosing until 32 hours after dosing
  Apparent total volume of distribution when dosed orally, based on the terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States